CLINICAL TRIAL: NCT00006773
Title: Phase I Evaluation of the Safety of PS 341 in the Treatment of Recurrent Gliomas
Brief Title: Bortezomib in Treating Patients With Recurrent Glioma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Administratively complete.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02367; NABTT-9910; U01CA062475 (NIH); CDR0000068326 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2000-12-06; First posted 2003-01-27 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Adult Anaplastic Astrocytoma; Adult Anaplastic Oligodendroglioma; Adult Giant Cell Glioblastoma; Adult Glioblastoma; Adult Gliosarcoma; Recurrent Adult Brain Tumor
MeSH Terms: conditions — Astrocytoma; Oligodendroglioma; Glioblastoma; Gliosarcoma; Brain Neoplasms | interventions — Bortezomib

ARMS (1):
- Treatment (bortezomib) (Experimental): Patients receive bortezomib IV over 3-5 seconds twice weekly for 2 weeks. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: bortezomib

INTERVENTIONS:
Drug: bortezomib — Given IV
  Other Names: LDP 341; MLN341; VELCADE

SUMMARY:
Phase I trial to study the effectiveness of bortezomib in treating patients who have recurrent glioma. Bortezomib may stop the growth of tumor cells by blocking the enzymes necessary for tumor cell growth

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the maximum tolerated dose of bortezomib with or without anticonvulsant drugs known to be metabolized by the P450 hepatic enzyme complex in patients with recurrent glioma.

II. Determine the biologic activity of this drug by measuring proteasome 20S activity in these patients.

III. Determine the effects of hepatic enzyme-inducing drugs, such as anticonvulsants, on biologic activity of this drug in these patients.

OUTLINE: This is a dose-escalation, multicenter study. Patients are stratified according to concurrent anticonvulsant drug use (phenytoin, carbamazepine, phenobarbital, primidone, or felbamate vs gabapentin, lamotrigine, valproic acid, or no anticonvulsant drugs).

Patients receive bortezomib IV over 3-5 seconds twice weekly for 2 weeks. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of bortezomib until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, 10 additional patients are treated with bortezomib at the MTD. Patients are followed every 2 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed progressive or recurrent malignant glioma

  * Anaplastic astrocytoma
  * Anaplastic oligodendroglioma
  * Glioblastoma multiforme
* Prior low-grade gliomas that have progressed to high-grade after therapy allowed
* Measurable disease by MRI or CT scan
* Performance status - Karnofsky 60-100%
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Bilirubin no greater than 1.5 mg/dL
* Transaminases no greater than 4 times upper limit of normal
* Creatinine no greater than 1.7 mg/dL
* Mini mental score at least 15
* No concurrent serious infection or other medical illness that would preclude study participation
* No other malignancy within the past 5 years except curatively treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix or breast
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after study participation
* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas) and recovered
* No more than 1 prior chemotherapy regimen
* At least 3 months since prior radiotherapy and recovered
* No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2001-05; Primary Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of bortezomib defined as the dose level below that at which > 1 of 3-6 patients experience DLT | 3 weeks
  Graded using the CTC version 2.0.

SECONDARY OUTCOMES:
Biological effectiveness estimated using 20S proteosome activity | Up to 6 years
  Simple descriptive measures will be used to examine the association between biological effect and the probability of toxicity and response.
Frequency of toxicity, graded using the CTC version 2.0 | Up to 6 years
  The proportion of patients with serious or life threatening toxicities will be estimated along with 95% confidence intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Olson, Principal Investigator — New Approaches to Brain Tumor Therapy Consortium
Locations (1):
- New Approaches to Brain Tumor Therapy Consortium, Baltimore, Maryland, United States